CLINICAL TRIAL: NCT06712693
Title: Venting Effects on Speech Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-26765
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Each participant will be fit with the investigational devices under three conditions: Power dome, Vented dome, and Open dome. Participant will complete the same tests under each condition. All participants will complete the same conditions.
Masking Description: Participants will know they are being fit with hearing aid, but will not be told which vent size or dome they are being fit with for any of the tests. The investigator scoring the speech test will not know which vent size/dome participant is wearing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): All participants will be tested using all three types of domes: Power, Vented, Open.
  Interventions: Device: Phonak Audeo Infinio Hearing Aid

INTERVENTIONS:
Device: Phonak Audeo Infinio Hearing Aid — Receiver-In-Canal hearing aid type that is coupled with either a custom earmold or a dome.

SUMMARY:
This study aims to gather behavioral data on the effect of earmold venting on speech performance in noise with a new noise reduction feature.

ELIGIBILITY:
Subjects fulfilling all of the following inclusion criteria are eligible for the investigation:

* 18-85 years of age
* Experienced hearing aid users
* N3-N4 hearing loss
* Fluent in English; ability to read and write in English
* Able to complete complex tasks
* Willing and able to provide informed consent
* Available for the data collection period

The presence of any one of the following exclusion criteria will lead to the exclusion of the subject:

* Self-reported active ear-related pathology (otorrhea, dizziness, sudden hearing loss or worsening of hearing, otalgia)
* Visible deformity of the ear
* Chronic, severe tinnitus
* Unilateral hearing loss
* Cognitive impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
AZ Bio Sentences | 1 day
  Sentences will be presented at a pre-determined Signal-to-Noise Ratio (SNR). The SNR will be the same for all three conditions (Power dome, Vented dome, Open dome). Percent correct will be calculated for all conditions. A higher percentage indicates better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.